CLINICAL TRIAL: NCT04198272
Title: Impact Evaluation of CyberRwanda: a Digital Health Intervention for Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: Youth Development Labs, Inc dba YLabs (Other); Society for Family Health, Rwanda (Unknown)
Responsible Party: Principal Investigator, Sandra McCoy, Associate Professor in Residence, University of California, Berkeley
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-04-12145
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-02

CONDITIONS: Pregnancy in Adolescence; Adolescent Health; Health Services Accessibility
Keywords: Adolescent health; Unintended pregnancy; Global health; Access to contraceptives

STUDY DESIGN:
Intervention Model Description: 3-arm cluster randomized controlled trial, clusters are secondary schools in Rwanda
Who Masked: Outcomes Assessor
Masking Description: Data analysts will be blind to intervention/control attribution
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Facilitated (Experimental): Schools that are randomized to this arm will be exposed to all of the components in the self-service version in addition to peer facilitation of the CyberRwanda platform at CyberRwanda clubs.
  Interventions: Behavioral: CyberRwanda
- Self-service (Active Comparator): Schools that are randomized to this arm will be exposed to the following components of the intervention:
  * Self-guided access to the online CyberRwanda platform; and
  * Promotion of the CyberRwanda program through school launch events.
  Interventions: Behavioral: CyberRwanda
- Control (No Intervention): Schools in this arm will not receive any intervention.

INTERVENTIONS:
Behavioral: CyberRwanda — The CyberRwanda intervention consists of three primary components: 1. STORIES: The CyberRwanda curriculum empowers youth to learn about family planning and reproductive health and employment skills and to set goals for their futures through age-appropriate, interactive, digital and printed stories and activities. 2. LEARN: Q&As and videos related to family planning and reproductive health. 3. SHOP: Youth can directly purchase health products, including menstrual hygiene and contraceptive products (emergency contraception, condoms, and oral contraceptive pills) online. The online health facility finder tool links youth to health facilities for longer-acting methods. All participating pharmacies will be trained to give unbiased, nonjudgmental information and services.
  Arms: Facilitated; Self-service

SUMMARY:
This protocol describes an evaluation of the CyberRwanda program, a digital health tool designed with and for adolescents in Rwanda, with a focus on successful futures, broadly, and family planning and reproductive health, more specifically. CyberRwanda is a tablet-based system that provides information on family planning and reproductive health through a set of vignettes. The program also allows users to order and purchase contraceptives, with pick up at nearby participating pharmacies. The program will be implemented in schools in eight districts in Rwanda. The investigators will conduct a 3-arm, cluster, randomized controlled trial to evaluate the impact of CyberRwanda on three primary outcomes: uptake of a contraceptive method, initiation of childbearing, and HIV testing. The investigators will compare two implementation models (facilitated and self-service) to a control arm at the school (cluster) level. The study will enroll 60 schools (20 per arm) and 100 students per school, and follow students for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Attending a study school at baseline in secondary school levels S1 or S2;
* Between 12 and 19 years of age;
* If <18 years of age: Assent and parental consent to participate in the study;
* If ≥ 18 years of age, informed consent to participate in the study;
* Willingness to provide valid contact information for study follow-up purposes.

Exclusion Criteria:

-

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 6078 (Actual)
Dates: Start 2021-02-20 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Uptake of a modern contraceptive method | 24 months
  The proportion of female youth who report currently using a modern method of contraception at endline (24 months). The primary outcome is expressed as a binary variable, defined as female youth who are currently using a modern method of contraception at endline versus female youth who are not using a modern method of contraception.
Initiation of childbearing | 24 months
  The proportion of female youth who report having ever been pregnant at endline (24 months), regardless of the pregnancy outcome. This outcome is expressed as a binary variable, defined as female youth who report having ever been pregnant versus female youth who report never having been pregnant.
HIV testing | 24 months
  The proportion of youth who have ever had an HIV test at endline (24 months). This outcome is expressed as a binary variable, defined as youth who report having ever been tested for HIV versus youth who report never having tested for HIV.

SECONDARY OUTCOMES:
FPRH Knowledge: % of youth that understand the phases of a girl's menstrual cycle | 24 months
  The total number of youth who can correctly identify a woman's fertile period, divided by the total number of youth.
Behavioral Intentions: % of youth who intend to use a modern contraceptive method in the next 12 months | 24 months
  The total number of youth, disaggregated by sex, who are very confident or confident that they will use contraception in the 12 months divided by the total number of youth who anticipate that they will have sexual intercourse in the next 12 months.
Self-efficacy Contraceptive Use: % of adolescents who are confident that they could get their partner(s) to use contraceptives/condoms if they desired | 24 months
  The total number of youth who state that they agree or strongly agree that they feel confident that they can negotiate contraception and condom use with their partners, divided by the total number of youth.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra McCoy, PhD, Principal Investigator — UC Berkeley
Locations (2):
- Rwanda (2):
  - Society for Family Health, Kigali
  - Youth Development Labs, Kigali

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hemono R, Gatare E, Kayitesi L, Hunter LA, Packel L, Ippoliti N, Cerecero-Garcia D, Contreras-Loya D, Gadsden P, Bautista-Arredondo S, Sayinzoga F, Mugisha M, Bertozzi SM, Hope R, McCoy SI. Effect of a digital school-based intervention on adolescent family planning and reproductive health in Rwanda: a cluster-randomized trial. Nat Med. 2024 Nov;30(11):3121-3128. doi: 10.1038/s41591-024-03205-1. Epub 2024 Aug 23. PMID 39179855
- [Derived] Hemono R, Gatare E, Kayitesi L, Hunter LA, Kunesh J, Packel L, Hope R, McCoy SI. Measuring sexual behavior among in-school youth in Rwanda: a cross-sectional analysis of self-reported timing of first sex and correlates of early sexual debut. Ann Epidemiol. 2023 Jul;83:35-39.e1. doi: 10.1016/j.annepidem.2023.04.005. Epub 2023 Apr 14. PMID 37060934
- [Derived] Nolan C, Packel L, Hope R, Levine J, Baringer L, Gatare E, Umubyeyi A, Sayinzoga F, Mugisha M, Turatsinze J, Naganza A, Idelson L, Bertozzi S, McCoy S. Design and impact evaluation of a digital reproductive health program in Rwanda using a cluster randomized design: study protocol. BMC Public Health. 2020 Nov 13;20(1):1701. doi: 10.1186/s12889-020-09746-7. PMID 33187485
- See also: CyberRwanda analysis plan pre-registered on the Open Science Framework (May 2021) — https://osf.io/jmz4u